CLINICAL TRIAL: NCT02914288
Title: Prospective Observation for Serial Changes of Acute Intracranial Artery Dissection Using High Resolution MRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government); Bracco Corporate (Industry)
Responsible Party: Principal Investigator, Seung Chai Jung, MD. PhD., Asan Medical Center
Other Study IDs: ICD_02
Record Dates: First submitted 2016-09-07; First posted 2016-09-26 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Cerebral Arterial Diseases; Dissecting Aneurysm of Cerebral Artery; Intimal Dissection
MeSH Terms: conditions — Cerebral Arterial Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: High resolution magnetic resonance imaging for intracranial vessel walls — High resolution magnetic resonance imaging for intracranial vessel walls at initial (optional), 1 month, 3 month, 6 month (optional), and 12 month

SUMMARY:
Intracranial artery disease has been more detected with development of HR-MR. HR-MR can depict vascular wall directly and give us more information beyond the pre-existing imaging modalities such as digital subtraction angiography, magnetic resonance angiography, computed tomography angiography. Hence, HR-MR is considered to become promising imaging modality for intracranial artery disease and many studies have been published recently. However, there was not enough to differentiate various intracranial artery disease such as atherosclerosis, dissection, moyamoya disease, vasculitis, reversible vasoconstriction syndrome. In real clinical arena, intracranial artery disease is too difficult to diagnose and distinguish among the disease. Of the disease, usefulness of HR-MR has been consistently published in the detection and diagnosis of intracranial artery dissection recently. HR-MR seems to be the most important and reliable imaging method in intracranial artery dissection as of now. Therefore, intracranial artery dissection is necessary to study using HR-MR. Intracranial artery dissection is dynamic vascular pathology. The geometric change is the most common among intracranial artery disease. However, there was no report about the geometric change in HR-MR. The investigators acquired retrospective data about the natural course of intracranial artery dissection in HR-MR and are preparing for publishing an article. However, the data is not prospective and not intraindividual comparison. Therefore, reliability is not enough to convince the natural course. If the investigators got prospective and intraindividual data, definite natural course of intracranial artery dissection could be acquired and would be helpful to diagnose the dissection and differentiate from other vascular pathologies. The prospective longitudinal information from this study could guide us as the important map on the confusing HR-MR findings. The protocols for imaging are as follows: initial (optional), 1 month, 3 month, 6 month (optional), 12 month.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* acute intracranial artery dissection

Exclusion Criteria:

* angioplasty, or stenting,
* contraindication for MR imaging,
* Hypersensitivity to gadolinium based contrast media,
* Pregnant or lactating women,
* Renal condition : eGFR < 60, 6) Patients unable and/or unwilling to comply with treatment or study instructions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Acute intracranial artery dissection
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Five proportions (%) of dissection findings | 12 months
  Visual detection based on PACS system by obsevers: Presence or absence of each finding (intimal flap, double lumen, intramural hematoma, aneursymal dilatation, wall enhancement): Proportions (%)= number of patients with presence of each finding/ number of all patients
Three diameters (mm) of dissecting arterial segment and contralateral segment | 12 months
  Outer diameter, Inner luminal diameter, Normal diameter (mm) by measured semi-automatic in-house analysis software based on Image J
Wall measurement (mm2) of dissecting arterial segment and contralateral segment | 12 months
  Wall area by measured semi-automatic in-house analysis software based on Image J: Wall area (mm2)= Outer wall area - luminal area
Remodeling index of dissecting arterial segment and contralateral segment | 12 months
  Remodeling index= outer wall area of dissection segment / [(outer wall area of proximal normal looking segment + outer wall area of distal normal looking segment)/2]
Extent (mm) of dissecting arterial segment and contralateral segment | 12 months
  Length (mm) on curved multiplanar reconstructed images by measured semi-automatic in-house analysis software based on Image J

CONTACTS AND LOCATIONS:
Overall Officials: Seung Chai Jung, MD.,PhD., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Seoul, South Korea